CLINICAL TRIAL: NCT06739018
Title: Comparison of Anterior Segment and Corneal Parameters in Keratoconus and High Myopic Astigmatism Using Schiempflug Imaging
Brief Title: Anterior Segment and Corneal Parameters in Keratoconus and High Myopic Astigmatism Using Schiempflug Imaging
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Youstena Saied Waheb, DR, Assiut University
Other Study IDs: pentacam parameters compare
Record Dates: First submitted 2024-11-27; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Keratoconus; High Myopia
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- keratoconic group: patients with keratoconus
  Interventions: Other: pentacam scheimpflug tomography
- high myopic astigmatim group: patients with high myopic astigmatism
  Interventions: Other: pentacam scheimpflug tomography

INTERVENTIONS:
Other: pentacam scheimpflug tomography — Pentacam tomography is not radiation-based. It uses Scheimpflug imaging, which involves a rotating camera that captures multiple images of the anterior segment of the eye. The system employs light-based technology to measure the front and back surfaces of the cornea, along with the anterior chamber and lens, creating a 3D model of the anterior eye structures.
  it uses light instead of ionizing radiation (like X-rays), it is considered safe and non-invasive for routine use in ophthalmology.
  * It was used to assess 23 parameters from topographic maps and 15 parameters from Belin-Ambrosio enhanced ectasia (BAD) display maps.
  * Parameters included keratometry readings, anterior and posterior sagittal curvature, corneal thickness, anterior chamber volume, and several indices from the BAD display map.
  * These parameters were analyzed to discriminate between keratoconus and high myopic astigmatism using Receiver Operating Characteristic (ROC) curves for diagnostic accuracy.

SUMMARY:
The purpose of this study was to compare Scheimpflug corneal tomography findings in keratoconus and high myopic astigmatic eyes, as well as to establish the parameters distinguishing keratoconus from high myopic astigmatism.

DETAILED DESCRIPTION:
Keratoconus is a progressive, non-inflammatory corneal ecstatic disorder caused by alteration in the structure and organization of corneal collagen fibers. It results in uneven steepening of the cornea, resulting in irregular astigmatism that cannot be totally corrected with glasses, impairing the quality of life . However, in many cases, increased axial length adds to the myopic component of refractive error . Thereafter, keratoconus patients frequently have axial high myopia with irregular astigmatism . Furthermore, early diagnosis of keratoconus aids in the timely management of the condition, thus improving patients' quality of life. According to research, high myopia, in addition to the degree of astigmatism, is an alarming sign that requires further corneal assessment to rule out any corneal abnormalities such as keratoconus. Furthermore, keratoconus could be misdiagnosed as meridional amblyopia attributable to myopic astigmatism due to the lack of corneal tomography measurements . As a result, it is critical to evaluate all high myopia patients, particularly those considering refractive surgery, for high-risk corneas.

The criteria for diagnosing and classifying keratoconus are based on anterior corneal curvature data obtained using Placido-based corneal topography . Early alterations in eyes with keratoconus, however, have been found on the posterior corneal surface . Scheimpflug imaging uses a revolving Scheimpflug camera to determine the front and back surfaces of the cornea, hence measuring the overall thickness. Several studies have utilized Scheimpflug tomography to evaluate anterior segment parameters between normal eyes and eyes with keratoconus , but the utility of Scheimpflug imaging to distinguish between keratoconus and high myopic astigmatism has not been thoroughly examined.

ELIGIBILITY:
Inclusion Criteria:

* keratoconus patient
* virgin clear cornea with high myopic astigmatism
* normal cornea with high myopic astigmatism

Exclusion Criteria:

* patients had previous ocular surgery
* ocular diseases rather than keratoconus
* contact lens wearer
* corneal opacity and corneal dystrophy

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The population represents individuals either have keratoconus or high mopic astigmatism and fit the inclusion and exclusion criteria to ensure proper comparison of corneal parameters .
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
overall corneal mean difference thickness between keratoconus and mopc astigmatism | baseline
  Scheimpflug imaging uses a revolving Scheimpflug camera to determine the front and back surfaces of the cornea, hence measuring the overall corneal mean difference thickness between keratoconus and mopc astigmatism as regarding central anterior chamber depth

CONTACTS AND LOCATIONS:
Overall Officials: Momen Aly, lecturer, Study Director — Assiut University
Locations (2):
- Egypt (2):
  - Assiut university, Asyut, Asyut Governorate
  - Assiut university, Asyut

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zaabaar E, Kyei S, Parkson Brew MAA, Boadi-Kusi SB, Assiamah F, Asiedu K. The utility of measures of anterior segment parameters of a Pentacam Scheimpflug tomographer in discriminating high myopic astigmatism from keratoconus. PLoS One. 2021 Dec 2;16(12):e0260648. doi: 10.1371/journal.pone.0260648. eCollection 2021. PMID 34855828